CLINICAL TRIAL: NCT07063004
Title: Combined Effects of Bruegger's Exercises and Upper Thoracic Mobilizations Along With Standard Physical Therapy in Patients With Non-specific Neck Pain
Brief Title: Combined Effects of Bruegger's Exercises and Upper Thoracic Mobilizations in Patients With Non-specific Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/24/0159 Maryam
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Neck Pain
Keywords: Pain; Disability; Manual therapy
MeSH Terms: conditions — Neck Pain; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bruegger's Exercise and Upper Thoracic Mobilization (Experimental): Bruegger's Exercise: The position will be held for 10 second at first session and then there will be an increment of 2 seconds during each session.
  Upper Thoracic Mobilization: Upper thoracic (T1-T6) mobilization (Maitland mobilization (Grade I, II and III; PA glide) applied in prone lying position from via spinous process. Amount of treatment will be 3-4 mobilizations for a vertebra for 30 seconds approximately.
  Interventions: Other: Bruegger's Exercise and Upper Thoracic Mobilization
- Standard Physical Therapy (Active Comparator): * Isometric exercises will be done for flexors, extensors, rotators, and lateral flexors of the neck. Isometrically contracting working muscle for 5 seconds against patients own hand, which was placed in compliance with the working muscles, with a total of 10 repetitions.
  * Passive stretching will apply to Upper trapezius, Levator scapulae, Sternocleidomastoid, Scalene, Pectoralis major and minor muscle for 3-5 repetition 10 with 20-30 second hold. Intensity of exercise will be prescribed according to patient's tolerance level. Duration of stretch will 15 to 30 seconds, 3-5repetition and for 10 minutes.
  * Postero-anterior Maitland mobilization (Grade I & II) for C1-C2, Maitland lateral PA glide (Grade-III & IV) for C3-C6. Time of oscillations will be two or three oscillations in a second for one to two minutes.
  Interventions: Other: Standard Physical Therapy

INTERVENTIONS:
Other: Bruegger's Exercise and Upper Thoracic Mobilization — Bruegger's Exercise: The position will be held for 10 second at first session and then there will be an increment of 2 seconds during each session.
  Upper Thoracic Mobilization: Upper thoracic (T1-T6) mobilization (Maitland mobilization (Grade I, II and III; PA glide) applied in prone lying position from via spinous process. Amount of treatment will be 3-4 mobilizations for a vertebra for 30 seconds approximately.
  Arms: Bruegger's Exercise and Upper Thoracic Mobilization
Other: Standard Physical Therapy — Isometric exercises will be done for flexors, extensors, rotators, and lateral flexors of the neck. Isometrically contracting working muscle for 5 seconds against patients own hand, which was placed in compliance with the working muscles, with a total of 10 repetitions.
  Passive stretching will apply to Upper trapezius, Levator scapulae, Sternocleidomastoid, Scalene, Pectoralis major and minor muscle for 3-5 repetition 10 with 20-30 second hold. Intensity of exercise will be prescribed according to patient's tolerance level. Duration of stretch will 15 to 30 seconds, 3-5repetition and for 10 minutes.
  Postero-anterior Maitland mobilization (Grade I & II) for C1-C2, Maitland lateral PA glide (Grade-III & IV) for C3-C6. Time of oscillations will be two or three oscillations in a second for one to two minutes.
  Arms: Standard Physical Therapy

SUMMARY:
Neck pain is a multifactorial disease, and is a major problem in modern society. Patients with NCNP usually have alterations in cervical proprioception and PS. They may also develop symptoms such as dizziness or vertigo. A recently published study shows that patients with NCNP suffer greater sensations of stunning and lack of proprioception than patients with benign paroxysmal vertigo.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial and will be conducted on general population in Gujrat. Non-probability convenient sampling will be used to collect the data. Sample size of 48 subjects with age group between 25-45 years will be taken. Data will be collected from the patients having present complaint of Nonspecific Neck pain. Outcome measures will be taken using Numeric pain rating scale (NPRS) for pain, Neck disability index (NDI) for measuring disability and goniometer for range of motion (ROM). An informed consent will be taken. Subjects will be selected based on inclusion and exclusion criteria and will be equally divided into two groups by random number generator table. Both the Groups will receive standard physical therapy, while Group A will receive bruegger's exercises and Group B will receive Upper thoracic mobilization. Outcome measures will be measured at baseline then after 4 weeks(post). Data analysis will be done by SPSS version 21.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females between 25 and 45 years of age with nonspecific neck pain, and Current neck pain of at least 3 months duration.

Exclusion Criteria:

* Cervical radiculopathy, History of whiplash injury and surgery

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | upto 4 weeks
  Patient level of pain will be assessed using the NPRS scale. The NPRS was used to capture the patient's level of pain. Patients were asked to indicate the intensity of their current pain level using an 11-point scale, ranging from 0 (no pain) to 10 (worst pain imaginable).
Neck Disability Index (NDI) | upto 4 weeks
  Patient level of Disability will be assessed using NDI. The NDI is a self-report questionnaire with 10-items: pain intensity, personal care, lifting work, headaches, concentration, sleeping, driving, reading, and recreation. The response to each item is rated on a 6-point scale from 0 (no disability) to 5 (complete disability). The numeric responses for each item are summed for a total score ranging between 0 and 50; however, some evaluators have chosen to multiply the raw score by 2 and then report the NDI on a 0-100% Higher scores represent increased levels of disability.
Universal Goniometer (UG) | upto 4 weeks
  A large UG having 12-inch arms and full-circle plastic body will be used for measuring ACROM..It will be used to measure cervical AROM: flexion, extension, lateral flexion, and rotation.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical and Rehabilitation Center, Gujrat, Gujrat, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kazeminasab S, Nejadghaderi SA, Amiri P, Pourfathi H, Araj-Khodaei M, Sullman MJM, Kolahi AA, Safiri S. Neck pain: global epidemiology, trends and risk factors. BMC Musculoskelet Disord. 2022 Jan 3;23(1):26. doi: 10.1186/s12891-021-04957-4. PMID 34980079
- [Background] Bernal-Utrera C, Gonzalez-Gerez JJ, Anarte-Lazo E, Rodriguez-Blanco C. Manual therapy versus therapeutic exercise in non-specific chronic neck pain: a randomized controlled trial. Trials. 2020 Jul 28;21(1):682. doi: 10.1186/s13063-020-04610-w. PMID 32723399
- [Background] Fandim JV, Nitzsche R, Michaleff ZA, Pena Costa LO, Saragiotto B. The contemporary management of neck pain in adults. Pain Manag. 2021 Jan;11(1):75-87. doi: 10.2217/pmt-2020-0046. Epub 2020 Nov 25. PMID 33234017
- [Background] Joshi S, Balthillaya G, Neelapala YVR. Thoracic Posture and Mobility in Mechanical Neck Pain Population: A Review of the Literature. Asian Spine J. 2019 Jun 3;13(5):849-860. doi: 10.31616/asj.2018.0302. Print 2019 Oct. PMID 31154701
- [Background] Arsh A, Darain H, Iqbal M, Rahman MU, Ullah I, Khalid S. Effectiveness of manual therapy to the cervical spine with and without manual therapy to the upper thoracic spine in the management of non-specific neck pain; a randomized controlled trial. J Pak Med Assoc. 2020 Mar;70(3):399-403. doi: 10.5455/JPMA.300523. PMID 32207414
- [Background] SALWA SHENDY PD, EL-KHOZAMY PD. Effect of Upper Thoracic Mobilization on Chronic Mechanical Neck Pain. The Medical Journal of Cairo University. 2019;87(June):1449-57.
- [Background] Hidalgo B, Hall T, Bossert J, Dugeny A, Cagnie B, Pitance L. The efficacy of manual therapy and exercise for treating non-specific neck pain: A systematic review. J Back Musculoskelet Rehabil. 2017 Nov 6;30(6):1149-1169. doi: 10.3233/BMR-169615. PMID 28826164